CLINICAL TRIAL: NCT06434142
Title: Wear Assessment of Novel PEEK Telescopic Attachment for Implant Retained Mandibular Overdenture
Brief Title: Wear Assessment of Novel PEEK Telescopic Attachment for Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamada Zaki Mahross Atia (Other)
Responsible Party: Sponsor-Investigator, Hamada Zaki Mahross Atia, Assistant Professor, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 751/306
Record Dates: First submitted 2024-05-19; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Attachment Disorder; Stress Disorder
Keywords: Telescopic attachment; Attachment Wear; Zirconia
MeSH Terms: conditions — Stress Disorders, Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient with zirconia copy (Experimental): Group I (study group) was the group of patients with zirconia as a primary copings that attach to the abutment and PEEK as a secondary coping telescopic attachment that attaches to the fitting surface of the denture.
  Interventions: Procedure: implant overdenture
- patients with cobalt chromium (CoCr) as primary copings (Experimental): Group II (control group) was the group of patients with cobalt chromium (CoCr) as primary copings attached to the abutment and PEEK as a secondary coping's telescopic attachment attached to the fitting surface of the denture.
  Interventions: Procedure: implant overdenture

INTERVENTIONS:
Procedure: implant overdenture — Following the two-stage surgical protocol, two dental implant fixtures with a length of 10 mm and a diameter of 3.7 mm were inserted at the canine area of the mandibular alveolar ridge.

SUMMARY:
To assess the wear of Zirconia-PEEK versus cobalt-chromium-PEEK telescopic attachments for implant retained complete mandibular overdenture. The wear of Zirconia-PEEK telescopic attachments can affect the retention of implant retained complete mandibular overdenture.

DETAILED DESCRIPTION:
Twelve completely edentulous patients were randomly chosen for implant retained telescopic overdentures construction and divided into two groups, where group I was a patient with zirconia copy, and group II was with cobalt chromium CoCr copy. The PEEK was constructed for both groups as a secondary coping telescopic attachment for the denture. The wear measurements of PEEK were performed optically by using a USB digital microscope with a built-in camera connected to a compatible personal computer at different intervals of baseline, 3, 6, and 9 months. The data was statistically analyzed and compared using student t-test, ANOVA, and Post Hoc Test.

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous
* free from any dental or systemic diseases

Exclusion Criteria:

* medically ill fit patient
* female patient

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-11 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
the mean wear values | at baseline
  measurement of the mean of wear between two test groups
the mean wear values | after 3 months interval
  measurement of the mean of wear between two test groups
the mean wear values | after 6 months interval
  measurement of the mean of wear between two test groups

CONTACTS AND LOCATIONS:
Locations (1):
- Hamada Zaki Mahross, Cairo, Egypt